CLINICAL TRIAL: NCT05643001
Title: Precision Clinical and Genetic Tools for Brain Health in Hemorrhagic Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Boston University (Other); Tufts University (Other)
Responsible Party: Principal Investigator, Christopher D. Anderson, MD, MMSc, Division Chief of Stroke and Cerebrovascular Disease, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2021P001597
Record Dates: First submitted 2022-11-30; First posted 2022-12-08 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2024-05

CONDITIONS: Hemorrhagic Stroke
MeSH Terms: conditions — Hemorrhagic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Electronic Health Record Notification (Experimental): For eligible patients presenting with an acute hemorrhagic stroke, a recommendation to measure low-density lipoprotein (LDL) and glycated hemoglobin A1c (HbA1c) together with their last measurement dates will be displayed in the patient's electronic health record through a best practice alert (BPA). The alert will display for the patient's provider when they first open the patient's chart. The provider may accept the automatically generated orders for both measurements displayed in the BPA, may modify one or both of the orders, or choose to dismiss the BPA.
  For patients that follow-up with the out-patient stroke clinic and received the in-patient intervention, a second BPA will suggest referrals to sleep study and audiology. The alert will display for the patient's provider when they first open the patient's chart. The provider may accept one or both of the referrals suggested by the BPA, or may choose to dismiss the BPA.
  Interventions: Other: In-patient and out-patient electronic health record alert

INTERVENTIONS:
Other: In-patient and out-patient electronic health record alert — Electronic health record best practice alert which suggests measurement of LDL and HbA1c (in-patient) and referrals to sleep study and audiology (out-patient)

SUMMARY:
The overall goal of this study is to increase health care provider awareness for common risk factors and comorbidities in patients with hemorrhagic stroke that are related to impaired brain health, to ultimately improve patients management and associated outcomes. The specific objective is to test the performance and effectiveness of a custom electronic health record (EHR)-based notification module at time of index hospitalization and at follow-up for hemorrhagic stroke survivors, before disparities in access to outpatient care may limit opportunities to intervene.

The investigators hypothesize that notification of health care providers through the EHR will increase measurements of low-density lipoprotein (LDL) and glycated hemoglogbin A1c (HbA1c) and increase evaluation and management rates for obstructive sleep apnea and hearing impairment.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older
* Presenting with a primary diagnosis of hemorrhagic stroke admitted to Massachusetts General Hospital inpatient stroke service

Exclusion Criteria:

* Patients not meeting above inclusion criteria
* Patients presenting with subdural or epidural hematoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2024-04-18 (Actual); Study Completion 2025-03-28 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with LDL measurements | 12 months
  Proportion of patients with any LDL measurements in the 12-months period surrounding acute hemorrhagic stroke (6-months before and 6-months follow-up following discharge). LDL measurements will be ascertained based on electronic health record documentation.
Proportion of patients with HbA1c measurements | 12 months
  Proportion of patients with any HbA1c measurements in the 12-months period surrounding acute hemorrhagic stroke (6-months before and 6-months follow-up following discharge). HbA1c measurements will be ascertained based on electronic health record documentation.

SECONDARY OUTCOMES:
Proportion of patients with management of obstructive sleep apnea | 6-months
  Proportion of patients with any attempt of management for obstructive sleep apnea (referral to a sleep specialist, sleep study, appointment at sleep specialist, new treatment for sleep apnea) in the 6-months period follow-up following discharge after acute hemorrhagic stroke. Management attempts will be ascertained based on electronic health record documentation among the patients for which the outpatient notification was displayed within this time period.
Proportion of patients with management of hearing impairment | 6-months
  Proportion of patients with any attempt of management for hearing impairment (referral for audiology, audiology, appointment at ENT, new hearing aids) in the 6-months period follow-up following discharge after acute hemorrhagic stroke. Management attempts will be ascertained based on electronic health record documentation among the patients for which the outpatient notification was displayed within this time period.
Proportion of patients with intensification of lipid-lowering therapy | 6-months
  Proportion of patients with prescription of a new lipid-lowering medication or increase in dose of an existing lipid-lowering medication in the 6-months period follow-up following discharge after acute hemorrhagic stroke. Medication prescriptions will be ascertained based on electronic health record documentation.
Proportion of patients with intensification of antidiabetic therapy | 6-months
  Proportion of patients with prescription of a new antidiabetic medication or increase in dose of an existing antidiabetic medication in the 6-months period follow-up following discharge after acute hemorrhagic stroke. Medication prescriptions will be ascertained based on electronic health record documentation.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher D Anderson, MD MMSc, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Prapiadou S, Tack RWP, Kimball TN, Mora S, Choksi D, Duperron MG, Senff JR, Kourkoulis C, Singh SD, Yechoor N, Parodi L, Tan BYQ, Rosand J, Mayerhofer E, Anderson CD. Enhancing Comorbidity Management in Patients With Hemorrhagic Stroke via an Electronic Health Record-Linked Best Practice Alert: A Pre/Post Study. J Am Heart Assoc. 2025 Dec 16;14(24):e042302. doi: 10.1161/JAHA.125.042302. Epub 2025 Dec 3. PMID 41334749